CLINICAL TRIAL: NCT05218720
Title: Association of Delirium and EuroSCORE II in Cardiac Surgery Patients
Brief Title: Delirium and EuroSCORE II in Cardiac Surgery
Status: Completed | Type: Observational
Sponsor: Aga Khan University (Other)
Responsible Party: Principal Investigator, Khalid Siddiqui, Assistant Professor, Aga Khan University
Other Study IDs: 2021-6153-19008
Record Dates: First submitted 2022-01-31; First posted 2022-02-01 (Actual); Last update posted 2023-07-27 (Actual); Status verified 2023-07

CONDITIONS: Delirium
Keywords: Cardiac Surgery; Post-operative Delirium; Coronary Artery Bypass Grafting; EuroSCORE II
MeSH Terms: conditions — Delirium; Emergence Delirium

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Diagnostic Test: EuroSCORE II — * Euro score II: Predicts risk of in-hospital mortality after major cardiac surgery. Risk category will be defined as very low risk <1, low risk 1-2.99, moderate risk 3-4.99, high risk >5.
  * CAM- ICU: The Confusion Assessment Method for the Intensive Care Unit (CAM-ICU) is a tool used to assess delirium among patients in the intensive care unit. It is an adaptation of the CAM which was originally developed to allow non-psychiatrists to assess delirium at the bedside. It ranges from 0 to 7, score greater to or equal to 3 will be considered positive for delirium, further categorized as 0-2 no delirium, 3-5 mild delirium 6-7 severe delirium with 7 being most severe.
  Other Names: CAM-ICU (The Confusion Assessment Method for the Intensive Care Unit)

SUMMARY:
Recognition of the delirium can be helped with delirium rating scales and checklists but mostly is a clinical diagnosis. It is important to recognize the large number of risk factors that can be associated with the condition but more importantly the type of surgery can also impact the development of post-operative dementia. In CABG (Coronary Artery Bypass Grafting) the overall incidence of POD(Post Operative Delirium) was 7.9% while it was 11.2% after valvular surgery according to one study.

Patients undergoing cardiac surgery mostly require risk stratification and prediction models are important tools for making medical decisions. One of the most used prediction models is the EuroSCORE risk model, which includes 17 independent variables and considers 30 days' operative mortality. It is used for assessing the risk associated with heart surgery and is based on the European cardiac surgical database.

The investigators will study the association between EuroSCORE II and delirium in cardiac surgery patients and see if an increased Euro score II association leads to the development of delirium.

DETAILED DESCRIPTION:
Patients undergoing cardiac surgery are at risk of developing delirium which is a frequent psychiatric condition found in ICU participants especially cardiac surgery patients. It presents with decreased levels of consciousness followed by a cognitive decline which is sometimes difficult to recognize along with altered sleep patterns. Hospital stay is increased for these patients, along with increased ICU stay which impacts morbidity and mortality and increases costs. The condition negatively impacts the post-op rehabilitation, quality of life and leads to social dependence for the patient, especially those who are older are at higher risks for long term cognitive dysfunction.

The diagnosis and monitoring of delirium remains a challenge because of the fluctuating course and different manifestations of the condition. There are wide variations in the incidence rates that are reported and are dependent on the diagnostic methods. The incidence of postoperative delirium in cardiac patients has been reported to be around 10-60 % and cognitive dysfunction occurs in up to 79% of these patients. Older patients have a high risk of developing deliriums in up to 73% of patients and in the ICU setting this rate is even higher up to 81%. Recognition of the disease can be helped with delirium rating scales and checklists but mostly is a clinical diagnosis. It is important to recognize the large number of risk factors that can be associated with the condition but more importantly the type of surgery can also impact the development of post-operative dementia. In CABG(Coronary Artery Bypass Grafting) the overall incidence of POD (Post Operative Delirium) was 7.9% while it was 11.2% after valvular surgery according to one study.

Patients undergoing cardiac surgery mostly require risk stratification and prediction models which are important tools for making medical decisions. One of the most used prediction models is the EuroSCORE II risk model, which includes 17 independent variables and considers 30 days' operative mortality. It is used for assessing the risk associated with heart surgery and is based on the European cardiac surgical database. Various studies have reported an association between higher scores on the EuroSCORE II system and the association with developing delirium.

With this, the investigators will study the association between EuroSCORE II and delirium in cardiac surgery patients and see if an increased preoperative EuroSCORE II leads to the development of delirium. It will help refute claims of the advantage of EuroSCORE II in predicting delirium after cardiac surgery. No such study has been performed in our country previously.

The rationale of this study is to see whether both the development of delirium and EuroSCORE II are independent of each other or if there is an association between the two.

ELIGIBILITY:
Inclusion Criteria:

* Age more than 18 years, both genders
* ASA I -IV, who will undergo elective cardiac surgeries (CABG, MVR, AVR), receiving invasive ventilation, at Aga Khan University Hospital.

Exclusion Criteria:

* Patients undergoing emergency cardiac surgeries
* Patients with a history of stroke within 6 weeks
* Patients with a previous history of delirium
* Patients with a previous history of psychiatric illness
* Patients with a history of medications for psychiatric illness
* Patients undergoing reopen surgeries

Ages: 18 Years to 80 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Patients (18-80 years) undergoing elective cardiac surgeries (CABG, MVR, AVR), receiving invasive ventilation
Sampling Method: Non-Probability Sample
Enrollment: 100 (Actual)
Dates: Start 2022-03-01 (Actual); Primary Completion 2023-05-23 (Actual); Study Completion 2023-05-23 (Actual)

PRIMARY OUTCOMES:
Incidence of delirium | Day 1
  An abrupt change in the brain that causes mental confusion and emotional disruption. According to DSM 5 criteria delirium is an acute condition. Signs and symptoms of delirium usually begin over a few hours or a few days. Delirium will be assessed by CAM-ICU score.

CONTACTS AND LOCATIONS:
Locations (1):
- Aga Khan University Hospital, Karachi, Sindh, Pakistan

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Norkiene I, Ringaitiene D, Kuzminskaite V, Sipylaite J. Incidence and risk factors of early delirium after cardiac surgery. Biomed Res Int. 2013;2013:323491. doi: 10.1155/2013/323491. Epub 2013 Sep 12. PMID 24102052
- [Background] Norkiene I, Ringaitiene D, Misiuriene I, Samalavicius R, Bubulis R, Baublys A, Uzdavinys G. Incidence and precipitating factors of delirium after coronary artery bypass grafting. Scand Cardiovasc J. 2007 Jun;41(3):180-5. doi: 10.1080/14017430701302490. PMID 17487768
- [Background] Koster S, Oosterveld FG, Hensens AG, Wijma A, van der Palen J. Delirium after cardiac surgery and predictive validity of a risk checklist. Ann Thorac Surg. 2008 Dec;86(6):1883-7. doi: 10.1016/j.athoracsur.2008.08.020. PMID 19022003
- [Background] Theologou S, Giakoumidakis K, Charitos C. Perioperative predictors of delirium and incidence factors in adult patients post cardiac surgery. Pragmat Obs Res. 2018 May 8;9:11-19. doi: 10.2147/POR.S157909. eCollection 2018. PMID 29773957
- [Background] European Delirium Association; American Delirium Society. The DSM-5 criteria, level of arousal and delirium diagnosis: inclusiveness is safer. BMC Med. 2014 Oct 8;12:141. doi: 10.1186/s12916-014-0141-2. PMID 25300023